CLINICAL TRIAL: NCT04369625
Title: Cross-sector Care for Children and Adolescents With Mentally Ill and Addicted Parents - Children of Mentally Ill Parents -Network - CHIMPS-NET
Brief Title: Children of Mentally Ill Parents-Network - CHIMPS-NET
Acronym: CHIMPS-NET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Silke Wiegand-Grefe, Prof. Dr. (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); Charite University, Berlin, Germany (Other); University Medical Center Rostock (Other); Immanuel Klinik Rüdersdorf (Unknown); Evangelisches Klinikum Bethel (Unknown); Universitätsklinikum Köln (Other); University of Göttingen (Other); Ruhr University of Bochum (Other); University Hospital Tuebingen (Other); University Hospital Freiburg (Other); Josefinum Augsburg (Unknown); University Hospital Augsburg (Other); Klinikum der Universität München (Unknown); University Hospital, Saarland (Other); University of Magdeburg (Other); Helios Kliniken Schwerin (Other); Universitätsklinikum Marburg (Unknown); Universitätsklinikum Koblenz - Landau (Unknown); Pfalzklinikum (Unknown); HELIOS Hospital, Erfurt, Germany (Other); Bezirkskrankenhaus Günzburg (Unknown); DAK Gesundheit (Other); Techniker Krankenkasse (Other); BARMER (Other); BKK Mobil Oil (Industry); KKH Kaufmännische Krankenkasse (Unknown); IKK Classic Krankenkasse (Unknown); AOK Hessen (Industry); University of Ulm (Other); University Hospital Heidelberg (Other); aQua-Institut (Unknown); Leibniz Universität, Center for Health Economics Research Hannover (Unknown); AFET Bundesverband für Erziehungshilfe e.V. (Unknown); Dachverband Gemeindepsychiatrie (Unknown); AOK Baden-Württemberg (Industry); LWL Klinik Gütersloh (Unknown); Staedtisches Klinikum Karlsruhe (Other)
Responsible Party: Sponsor-Investigator, Silke Wiegand-Grefe, Prof. Dr., Prof. Dr., Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: U1111-1244-6111
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Mental Health Issue
Keywords: children of mentally ill parents; e-mental health; early detection and early treatment of mental disorders

STUDY DESIGN:
Intervention Model Description: Each of the four interventions will be evaluated in a separate prospective, randomized-controlled trial (RCT); overall, four randomized-controlled trials will be performed. Each of the four control groups receive treatment as usual (TAU). Each of the four studies will include two groups: one intervention group (IG) and one control group (TAU), i.e. CHIMPS-T vs. KG (TAU), CHIMPS-MFT-group vs. KG (TAU), CHIMPs-P vs. KG (TAU), iCHIMPS vs. KG (TAU).
Who Masked: Investigator
Masking Description: Assessors are blind regarding the randomization (group affiliation) of the families.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CHIMPS-T (Experimental): (Children of mentally ill parents) is a family-oriented lowfrequency brief therapy for diagnosis and treatment of mental disorders in children and adolescents. CHIMPS-T is based on a theory model, needs analyses and the pioneering studies of Williams Beardslee. The CHIMPS approach was tested, evaluated and manualized in an initial project (2007-2011).
  Interventions: Behavioral: CHIMPS-T
- CHIMPS-P (Experimental): CHIMPS-P is a family-oriented prevention for children and adolescents without signs of mental disorders in the initial screening. These families will receive the 3 family sessions from the modular CHIMPS intervention. The sessions will be carried out by a social worker (based on the Finnish model "Let's talk about children (Solantaus), but in a family setting "Let's talk WITH children").
  Interventions: Behavioral: CHIMPS-P
- The CHIMPS-MFT-group (Experimental): The CHIMPS-MFT-group is a prevention with a multi-family setting based on the CHIMPS approach. The multi-family intervention comprises 8 sessions for children and adolescents without psychiatric disorders and their families: preliminary talk, one additional session with the family (if needed), multifamily group with three to six other families, concluding session.
  Interventions: Behavioral: CHIMPS-MFT-group
- iCHIMPS (Experimental): iCHIMPS is an online intervention. In terms of content, iCHIMPS is based on the CHIMPS program as well as on other evidence-based interventions of the study group. iCHIMPS will also be comprised of one module for children and adolescents as well as one module for parents; moreover; modules for the family system will be included. Overall, 8 consecutive online modules as well as elective modules will be included. These modules (e.g., dealing with difficult situations, emotion regulation, taboos and shame, self-worth) will be provided based on the specific constellation of children and adolescents of mentally ill parents. iCHIMPS will be completed by 2 booster session within a six months follow-up.
  Interventions: Behavioral: iCHIMPS
- Treatment as usual (No Intervention): The treatment as usual implies that families of the control group receive the treatment that is customary in regular care. Thus, these families normally don't receive any post-treatment. If, however, a member of a control group family appears to have an urgent need for treatment (every family receives a comprehensive diagnostic investigation at the beginning of the study), the respective family will be placed in the ambulatory care system.

INTERVENTIONS:
Behavioral: CHIMPS-T — CHIMPS-T (Children of mentally ill parents) is a family-oriented lowfrequency brief therapy for diagnosis and treatment of mental disorders in children and adolescents.
  Arms: CHIMPS-T
Behavioral: CHIMPS-P — CHIMPS-P is a family-oriented prevention for children and adolescents without signs of mental disorders in the initial screening. These families will receive the 3 family sessions from the modular CHIMPS intervention.
  Arms: CHIMPS-P
Behavioral: CHIMPS-MFT-group — The CHIMPS-MFT-group is a prevention with a multi-family setting based on the CHIMPS approach. The multi-family intervention comprises 8 sessions for children and adolescents without psychiatric disorders and their families.
  Arms: The CHIMPS-MFT-group
Behavioral: iCHIMPS — iCHIMPS is an online intervention. In terms of content, iCHIMPS is based on the CHIMPS program as well as on other evidence-based interventions of the study group. iCHIMPS will also be comprised of one module for children and adolescents as well as one module for parents; moreover; modules for the family system will be included.
  Arms: iCHIMPS

SUMMARY:
In order to identify psychological stress in children and adolescents of mentally ill parents as early as possible, four special intervention programs (CHIMPS-therapy, CHIMPS-Prevention-single, CHIMPS-MFT-group, iCHIMPS) have been developed. These four intervention programs are based on the initial medical situation, indication and need of the families. Thereby, an individually tailored counseling service will be provided. With this current project, the four counseling approaches will be tested at 19 study sites in 12 federal states in Germany. Moreover, the interventions long-term efficacy will be evaluated.

DETAILED DESCRIPTION:
The central objectives of the study at hand are the implementation, evaluation and transfer of three evidence-based innovative forms of care (CHIMPS-Therapy, CHIMPS-MFT-Group, CHIMPS-Prevention-Single) for children and adolescents (aged 3 to 18 years) with mentally ill parents at the 19 participating study cites in 12 federal states of Germany. In addition, iCHIMPS, an online intervention based on the CHIMPS concept for the whole family, will be developed.

The four innovative forms of care include diagnostic, prevention and - if needed - therapy in order to treat psychological symptoms of children and adolescents as early as possible. Thereby, chronification will be prevented and the cycle of transgenerational transmissions of psychiatric disorders will be broken. Each of the four interventions will be evaluated in a separate prospective, randomized-controlled trial (RCT); overall, four randomized-controlled trials will be performed. Each of the four control groups receives treatment as usual (TAU). Each of the four studies will include two groups: one intervention group (IG) and one control group (KG), i.e. CHIMPS-T vs. KG (TAU), CHIMPS-MFT-group vs. KG (TAU), CHIMPs-P vs. KG (TAU), iCHIMPS vs. KG (TAU). Central psychosocial outcomes will be assessed at four time points (t1, t2, t3, t4) at baseline as well as after six, 12 and 18 months. Due to a longer development period, iCHIMPS will have three times of measurement over a period of nine months (baseline, post-intervention after 2 months as well as six-months-followup) within the project term. Outcomes will be assessed from the perspectives of the mentally ill parent, the partner (if available), every child and adolescent (0 - 9 years only external assessment; from 10 years of age additional self-assessment) and the professionals. A special characteristic of the study at hand is the comprehensive accompanying evaluation of medical biometry, health economics and qualitative evaluation.

In addition, various sub-projects for systematic implementation will be conducted:

optimization of pathway to care, knowledge and skills of professionals, development of a screening instrument and external quality assurance. In order to evaluate the effect of these three implementation strategies, an implementation study with a cluster-randomized trial was designed. Nineteen clinical centers are taking part in the implementation study. Nine of the nineteen clinical centers will receive the support of one of the three implementation strategies, the other ten clinical centers make up the control group and do not get a specific implementation support. The allocation is randomized. With three questionnaires in the investigator's implementation study we want to identify factors hindering or promoting implementation processes.

ELIGIBILITY:
Inclusion Criteria:

1. Familiy with at least one psychiatrically ill parent (all F-diagnoses in ICD-10) and at least one child between the age of 3 and 18 years.
2. Consent to participate in the study.
3. Sufficient knowledge of the German language of parents and children.
4. Consent to data processing of the insurance companies, if insured with one of the participating insurance companies.
5. Consent to participation in special care (in case of interventions).

Exclusion Criteria:

Severe psychiatric disorders and impairments of parents or children with acute symptoms such as suicidal tendencies, severe depression, addictions, acute psychotic symptoms etc., which will not be sufficiently supplied by these new lowfrequency interventions.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 858 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Children's and adolescent's psychiatric symptomatology (CBCL) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Children's and adolescent's psychiatric symptomatology, assessed from the perspective of the parents by the Child Behaviour Checklist (CBCL 1,5-5; Achenbach & Rescorla, 2000), (CBCL 6-18R; Döpfner, Pflück, Kinnen, & Arbeitsgruppe Deutsche Child Behavior Checklist, 2014).

SECONDARY OUTCOMES:
Sociodemographic information | At baseline of the study]
  Sociodemographic information of the parents, assessed from the perspective of the parents.
Psychiatric disorders of the children and adolescents (YSR) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Psychiatric disorders of the children and adolescents, assessed from the perspective of the parents by the "Youth Self Report" (YSR; Döpfner, Pflück, Kinnen & Arbeitsgruppe Deutsche Child Behavior Checklist, 2014).
Psychiatric disorders of the children and adolescents (K-SADS-PL) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Psychiatric disorders of the children and adolescents, assessed from the perspective of an external rater by the Kiddie-SADS (K-SADS-PL) (Delmo, Weiffenbach, Gabriel, Stadler & Poustka, 2001).
Psychiatric symptomatology of the children and adolescents (GAF) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Psychiatric symptomatology of the children and adolescents, assessed from the perspective of an external rater by the "Global Assessment of Functioning" (GAF; Saß, Wittchen, Zaudig & Houben, 2003).
Mental health of the parents (BSI) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Mental health of the parents, assessed from the perspective of the parents by the "Brief Symptom Inventory" (BSI; Franke, 2000).
Mental health of the parents (PHQ) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Mental health of the parents, Mental health of the parents, assessed from the perspective of the parents by the "Patient Health Questionnaire" (PHQ; PHQ; Löwe, Spitzer, Zipfel & Herzog, 2002).
Mental health of the parents (GAF) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Mental health of the parents, assessed from the perspective of an external rater by the "Global Assessment of Functioning" (GAF; Saß, Wittchen, Zaudig & Houben, 2003).
General anxiety of the parents (GAD-7) | Change from baseline of the study at 6,12 and 18 months after the randomization
  General anxiety of the parents, assessed from the perspective of the parents by the "Gerneralized Anxiety Disorder-7" (GAD-7; Kroenke, Spitzer, Williams, Monahan, & Löwe, 2007).
Health-related quality of life of the parents (SF-12) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Health-related quality of life of the parents, assessed from the perspective of the parents by the "Short Form 12" (SF-12; Bullinger & Kirchberger, 1998)
Health-related quality of life of the parents (EQ-5D) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Health-related quality of life of the parents, assessed from the perspective of the parents by the EQ-5D (EQ-5D; Brooks, Rabin & Charro, 2003; Hinz, Klaiberg, Brahler & Konig, 2006).
Health-related quality of life of the children and adolescents (KIDSCREEN) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Health-related quality of life of the children and adolescents, assessed from the perspective of the child/adolescent (from 10 years of age) and from the perspective of the parents by the Kidscreen-27 (The KIDSCREEN Group Europe, 2006).
Family functioning (GARF) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Family functioning, assessed from the perspective of an external rater by the "Global Assessment of Relational Functioning" (GARF; Saß, Wittchen, Zaudig & Houben, 2003).
Family functioning (FB-A) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Family functioning, assessed from the perspective of the parents and the children and adolescents (from 10 years of age) by the "Allgemeiner Familienfragebogen" (FB-A; Cierpka & Frevert, 1995)
Social support of the parents (OSSQ) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Social support of the parents, of the children and adolescents, assessed from the perspective of the parents, of the children and adolescents (from 10 years of age) by the "Oslo Social Support Questionnaire" (OSSQ; Dalgard, 2006).
Parental stress coping (EBI) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Parental stress coping, assessed from the perspective of the parents by the "Elterliches Belastungsinventar" (EBI; Tröster, 2010).
Treatment evaluation (FBB) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Treatment evaluation, assessed from the perspective of the parents, the children and adolescents (from 10 years of age) as well as from the therapist by the "Fragebogen zur Behandlungsbeurteilung" (FBB; Mattejat & Remschmidt, 1999).
Satisfaction with the treatment (ZUF-8) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Satisfaction with the treatment of the parents, of the children and adolescents, assessed from the perspective of the parents and from the perspective of the children/adolescents (from 10 years of age) by the "ZUF-8" (Schmidt, Lamprecht & Wittmann, 1989).
Therapeutic activity and therapeutic processes (VPPS) | During the intervention
  Therapeutic activity and therapeutic processes, assessed from the perspective of the therapist by the "Vergleichende Psychotherapy Prozess Skalen" (VPPS; Beutel et al., 2016).
Treatment costs (CAMHSRI-DE) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Treatment costs of the children and adolescents, assessed from the perspective of an external rater by the German version of the "Children and adolescent mental health services receipt inventory" (CAMHSRI-DE; Kilian, Losert, McDaid, Park, Knapp, Beecham, Kusakovskaja, Murauskiene & the CAMHEE Project, 2009).
Treatment costs (CSSRI-DE) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Treatment costs of the parents, assessed from the perspective of an external rater by the German version of the "Client Socioeconomic and Services Receipt Inventory" (CSSRI-DE; Roick, Kilian, Matschinger, Bernert, Mory & Angermeyer, 2001).
Family-oriented attitude (FFMHPQ) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Family-oriented attitude, assessed from the clinical employee's point of view by the German version of the "Family Focused Mental Health Practice Questionnaire" (FFMHPQ, Laser et al., 2019).
Implementation components (ICQ) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Implementation components, assessed from the clinical employee's point of view by the German version of the "Implementation Components Questionnaire" (ICQ, Laser, Skogøy, Maybery & Wiegand-Grefe, 2019).
Implementation Satisfaction (ISS) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Implementation Satisfaction, assessed from the clinical employee's point of view by the German version of the "Implementation Satisfaction Scale" (ISS, Laser, Skogøy, Maybery & Wiegand-Grefe, 2019).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Universitätsklinikum Hamburg-Eppendorf, Klinik für Kinder- und Jugendmedizin, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Derived] Laser C, Pawils S, Daubmann A, Zapf A, Wiegand-Grefe S. Different perspectives in psychiatry: how family-oriented are professionals in Germany? BMC Psychiatry. 2024 Feb 20;24(1):142. doi: 10.1186/s12888-024-05562-0. PMID 38378503
- [Derived] Laser C, Modarressi A, Skogoy BE, Reupert A, Daubmann A, Holler A, Zapf A, Pawils S, Taubner S, Winter S, Maybery D, Wiegand-Grefe S. Clinical Implementation and Evaluation of Three Implementation Interventions for a Family-Oriented Care for Children of Mentally Ill Parents (ci-chimps): Study Protocol for a Randomized Controlled Multicenter Trial. Front Psychiatry. 2022 Feb 28;13:823186. doi: 10.3389/fpsyt.2022.823186. eCollection 2022. PMID 35295776